CLINICAL TRIAL: NCT03360487
Title: Effect of Photobiomodulation Treatment in the Sublingual Region and Along the Spinal Column in Individuals With Multiple Sclerosis: Protocol for a Randomized, Controlled, Double-blind, Clinical Trial
Brief Title: Effect of Photobiomodulation Treatment in Individuals With Multiple Sclerosis:
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FBMEM
Record Dates: First submitted 2017-11-17; First posted 2017-12-04 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sham photobiomodulation in the sublingual region (Sham Comparator): A disposable plastic wrap will cover the application pen for the purposes of hygiene, and the laser will be placed for 10 minutes, without being turned on.
  Interventions: Radiation: Photobiomodulation in the sublingual region
- Photobiomodulation in the sublingual region (Active Comparator): A disposable plastic wrap will cover the application pen for the purposes of hygiene, and the region will be irradiated for 10 minutes.
  Interventions: Radiation: Photobiomodulation in the sublingual region
- Sham photobiomodulation along the spinal cord (Sham Comparator): Transcutaneous irradiation of the spinal cord will be pretended on segments corresponding to the nerve roots of the lumbosacral plexus (T12-S5) and cervicothoracic plexus (C5-T1-2). Twenty points will be wakely irradiated for 30 seconds (total treatment time: 10 minutes).
  Interventions: Radiation: Photobiomodulation in the spinal cord
- Photobiomodulation along the spinal cord (Active Comparator): Transcutaneous irradiation of the spinal cord will be performed on segments corresponding to the nerve roots of the lumbosacral plexus (T12-S5) and cervicothoracic plexus (C5-T1-2). Twenty points will be irradiated for 30 seconds (total treatment time: 10 minutes).
  Interventions: Radiation: Photobiomodulation in the spinal cord
- Sham Photobiomodulation in the radial artery (Sham Comparator): Intravascular laser irradiation will be applied to the skin in the region of the radial artery with a specific turned-off bracelet of the DMC laser Therapy EC model.
  Interventions: Radiation: Photobiomodulation in the radial artery
- Photobiomodulation in the radial artery (Active Comparator): Intravascular laser irradiation will be applied to the skin in the region of the radial artery with a specific bracelet of the DMC laser Therapy EC model.
  Interventions: Radiation: Photobiomodulation in the radial artery

INTERVENTIONS:
Radiation: Photobiomodulation in the sublingual region — In the group submitted to sublingual irradiation, disposable plastic wrap will cover the application pen for the purposes of hygiene, and irradiation will take 10 minutes.
  Arms: Photobiomodulation in the sublingual region; Sham photobiomodulation in the sublingual region
Radiation: Photobiomodulation in the spinal cord — Transcutaneous irradiation of the spinal cord will be performed on segments corresponding to the nerve roots of the lumbosacral plexus (T12-S5) and cervicothoracic plexus (C5-T1-2). Twenty points will be irradiated for 30 seconds (total treatment time: 10 minutes).
  Arms: Photobiomodulation along the spinal cord; Sham photobiomodulation along the spinal cord
Radiation: Photobiomodulation in the radial artery — Intravascular laser irradiation will be applied to the skin in the region of the radial artery with a specific bracelet of the DMC laser Therapy EC model.
  Arms: Photobiomodulation in the radial artery; Sham Photobiomodulation in the radial artery

SUMMARY:
Background: Multiple sclerosis (MS) is an autoimmune disease, for which the forms of treatment are medication and rehabilitation. However, in vitro and in vivo studies have demonstrated that photobiomodulation can be an effective treatment modality for inflammatory diseases, including MS. Photobiomodulation has a broad range of benefits, such as the avoidance of cell and tissue death, the stimulation of healing and injury repair, reductions in pain, edema and inflammation, cell proliferation and even apoptosis. The outcomes of photobiomodulation include the regeneration of cells, the stimulation of the growth of Schwann cells, a reduction in spasticity, functional improvements, a reduction in nitric oxide levels and the upregulation of the cytokine IL10, demonstrating that this therapeutic modality can offer neuro-protection.

Methods: A randomized, controlled, double-blind, clinical trial is proposed. The patients will be divided into six groups. Groups 1 and 2 will receive sham and active photobiomodulation in the sublingual region, respectively. Groups 3 and 4 will receive sham and active photobiomodulation along the spinal cord, respectively. Group 5 will receive placebo treatment with photobiomodulation on the skin in the region of the radial artery with a specific bracelet. Group 6 will be treated with photobiomodulation on the skin in the region of the radial artery with a specific bracelet.

Discussion: Treatment for MS is directed at the immune response and slowing the progression of the disease. This is one of the first clinical trials with sublingual and along the spinal cord photobiomodulation, which could help establish a new, promising treatment of the disease associated with pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS;
* Age between 18 and 60 years;
* Currently undergoing pharmacological treatment;
* Capable of understanding and following verbal instructions;
* score of < 7 on the Expanded Disability Status Scale;
* No restriction will be imposed regarding gender.

Exclusion Criteria:

* Other autoimmune diseases;
* Neoplasias;
* Heart failure;
* Respiratory failure;
* Renal insufficiency;
* Hepatic insufficiency;
* Acquired immunodeficiency syndrome;
* Patients with relapses of the disease will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress | Through study completion, about one year.
  The concentration of endogenous nitrite will be evaluated in serum samples using the Total Nitric Oxide and Nitrate/Nitrite Parameter Assay Kit (R&D) according to the manufacturer´s instructions. Briefly, 50 µL sample will be incubated in 96 well plates with the reaction diluent provided by the kit, Griess Reagent I and II for 10 min at room temperature. Reactions will be read at 540 nm.
Tumor Necrosis Factor Alpha | Through study completion, about one year.
  The quantification of the serum levels of IL-10 and TNFα will be performed using the Human IL-10 and THF-alpha ELISA MAX (Biolegend), according to the manufacturer's instructions. Briefly, plates will be coated with the capture anti-IL-10 or anti-TNF-alpha monoclonal antibody for 18h at 8°C, washed and then incubated with the reagent provided by the kit to block non-specific binding and to reduce background. Samples will be added to each well at room temperature for 2h and after wash, detection antibody solution will be added. Reactions will be revealed with the Avidin-HRP solution and the absorbance will be read at 450nm.
Interleukin-10 | Through study completion, about one year.
  The quantification of the serum levels of IL-10 and TNFα will be performed using the Human IL-10 and THF-alpha ELISA MAX (Biolegend), according to the manufacturer's instructions. Briefly, plates will be coated with the capture anti-IL-10 or anti-TNF-alpha monoclonal antibody for 18h at 8°C, washed and then incubated with the reagent provided by the kit to block non-specific binding and to reduce background. Samples will be added to each well at room temperature for 2h and after wash, detection antibody solution will be added. Reactions will be revealed with the Avidin-HRP solution and the absorbance will be read at 450nm.

SECONDARY OUTCOMES:
EDSS | Through study completion, about one year.
  The participants will be evaluated before and after treatment using the Expanded Disability Status Scale administered by a physiotherapist.

CONTACTS AND LOCATIONS:
Locations (1):
- UNINOVE, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Silva T, Alencar RC, de Souza Silva BC, Viana ECOM, Fragoso YD, Gomes AO, Cristina Chavantes M, Deana AM, Gallo JMAS, Fernandes KPS, Mesquita-Ferrari RA, Bussadori SK. Effect of photobiomodulation on fatigue in individuals with relapsing-remitting multiple sclerosis: a pilot study. Lasers Med Sci. 2022 Oct;37(8):3107-3113. doi: 10.1007/s10103-022-03567-3. Epub 2022 May 2. PMID 35499744
- [Derived] Silva T, Fragoso YD, Destro Rodrigues MFS, Gomes AO, da Silva FC, Andreo L, Viana A, Teixeira da Silva DF, Chavantes MC, Tempestini Horliana ACR, De Angelis K, Deana AM, Branco LP, Santos Fernandes KP, Motta LJ, Mesquita-Ferrari RA, Bussadori SK. Effects of photobiomodulation on interleukin-10 and nitrites in individuals with relapsing-remitting multiple sclerosis - Randomized clinical trial. PLoS One. 2020 Apr 7;15(4):e0230551. doi: 10.1371/journal.pone.0230551. eCollection 2020. PMID 32255785